CLINICAL TRIAL: NCT01599065
Title: Comparison of a MAGNET Protocol Versus "off-on" Protocol for Patients With Implantable Cardioverter Defibrillators Undergoing Procedures Requiring Electrocautery
Brief Title: Comparison of a MAGNET Protocol Versus "off-on" Protocol for Patients With Implantable Cardioverter Defibrillators
Acronym: MAGNET
Status: Completed | Type: Observational
Sponsor: Midwest Heart Foundation (Other)
Collaborators: Abbott Medical Devices (Industry); Boston Scientific Corporation (Industry); Medtronic (Industry)
Responsible Party: Principal Investigator, Karen Larimer, PhD, Investigator, Midwest Heart Foundation
Other Study IDs: 01-2011
Record Dates: First submitted 2012-05-10; First posted 2012-05-15 (Estimated); Last update posted 2013-10-21 (Estimated); Status verified 2012-05

CONDITIONS: Sudden Cardiac Death; Arrhythmia; Heart Failure
Keywords: ICD; internal cardioverter defibrillator; electrocautery
MeSH Terms: conditions — Death, Sudden, Cardiac; Arrhythmias, Cardiac; Heart Failure | interventions — Magnets

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Magnet: group treated by disabling ICD during procedure
  Interventions: Other: Magnet or Off-On
- Off-On: Group having ICD turned off during the procedure
  Interventions: Other: Magnet or Off-On

INTERVENTIONS:
Other: Magnet or Off-On — Randomized to ICD suspension using a magnet or turning the ICD off and then back on.

SUMMARY:
The purpose of this study is to compare the two options for management of ICDs (internal cardioverter defibrillators) in patients undergoing procedures with electrocautery: (1) programming ICD therapies "off," or (2) use of a magnet to suspend ICD therapies By comparing these two techniques the investigators hope to demonstrate the efficiency of using an ICD magnet protocol during perioperative management of patients undergoing electrocautery procedures. Secondary purposes are to gain further information on health care resources, incidence of EMI, handoff communications and to document lack of adverse events in either group.

Primary objective will be: ICD therapy "off times" will be less with the use of a magnet protocol compared to an "off-on" protocol. Secondary objectives will be: (1) Healthcare resources (time and costs of skilled personnel) will be less using a magnet protocol compared to an off-on protocol, and (2) there will be no difference between adverse events in the magnet protocol compared to an off-on protocol. The incidence of EMI and number of handoff communications will be documented.

The investigators hypothesis is that the number of minutes with ICD therapies "off" will be significantly less with magnet use. The investigators also expect health care resources to be less with magnet use compared to reprogramming.

DETAILED DESCRIPTION:
The study design will be a prospective multi-center randomized controlled trial where subjects will be randomized to either a control group (ICD "off-on" group) or to the experimental group (magnet group) within blocks of type of procedure and site.

Subjects will be enrolled at the time of their procedure and will remain in the study until their post operative device interrogation. This could take place that same day ("off on" group or registry) or at their next ICD clinic visit or remote transmission (no more than 3 months from the procedure).

The study duration from first enrollment to closure is expected to last approximately 12 months. There will be only two enrolling centers and the target sample size is 150 subjects from various manufacturers. No specific sample size was calculated as this is a pilot study.

ELIGIBILITY:
Inclusion criteria

* Age > 18 years
* Have a pectorally implanted ICD
* Be scheduled for surgical procedure with anticipated electrocautery, OR
* Be scheduled for endoscopic procedure with anticipated electrocautery, OR
* Be scheduled for interventional radiology procedure with anticipated electrocautery
* Have a planned procedure with anticipated EC > 15 cm (6 in) from ICD generator*
* Have an ICD from the following manufacturer:

  * Medtronic, Inc., OR
  * Boston Scientific (formerly Guidant/CPI), OR
  * St. Jude Medical
* Be able to speak and understand English
* Be willing to sign consent form

  * While subjects having procedures < 15 cm (6 in) from generator will be excluded from the main study they will qualify to be placed in the registry.

Exclusion criteria

* Be scheduled for a surgical, endoscopic or radiologic procedure where electrocautery is not anticipated
* Be scheduled for a surgical, endoscopic or radiologic procedure where only bipolar electrocautery is planned (ophthalmologic procedures)
* Have an ICD from Boston Scientific under Product Advisory related to magnet performance.
* Have an ICD from the manufacturer ELA or Biotroniks

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have an ICD and are patients at Edward Hospital or Advocate Good Samaritan undergoing surgical, endoscopic and interventional radiologic procedures will be considered for the study. Hospital and cardiology practice staff will identify potential subjects by reviewing surgical, endoscopic and interventional radiologic procedure schedules. When patients with an ICD are identified research staff will be notified. Any scheduled adult patient with a past medical history of an ICD will be considered for participation. If electrocautery is anticipated for the procedure this patient will be screened for the study.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2011-12; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Number of minutes ICD therapy suspended will be less using a magnet protocol compared to number of minutes ICD therapy suspended using an "off-on" protocol. | Up to 90 days

SECONDARY OUTCOMES:
Healthcare resources will be less using a magnet protocol compared to an "off-on" protocol. Measures: Cost in dollars | Up to 90 days
  Cost of skilled personnel (cost is defined as number of minutes skilled personnel engaged in active management or waiting to be engaged in active management [and not otherwise productive] in management of subject) and cost of equipment (ie. transport monitor, defibrillator and pads) or any equipment necessary to man-age the subject that is unique to either magnet protocol or "off-on" protocol.
There will be no difference between adverse events using the magnet protocol compared to using an "off-on" protocol. | Up to 90 days
  1. proportion of subjects with arrhythmias requiring therapy
  2. proportion of subjects with inappropriate ICD therapies
  3. proportion of subjects with pacing inhibition
  4. proportion of subjects with magnet not secured during procedure
The incidence of EMI will be documented in relation to surgical locations: head/neck, thorax, abdomen/pelvis, upper extremity, lower extremity. | Up to 90 days
  Number of episodes of EMI
Number of handoff communication quantified. | Up to 90 days
  Handoff communications defined as "an exchange of information between staff regarding the ICD subject".

CONTACTS AND LOCATIONS:
Overall Officials: Janet Gifford, MSN, APN, Principal Investigator — Edward Hospital/Midwest Heart Foundation; Karen Larimer, PhD, ACNP, Principal Investigator — Midwest Heart Specialists-Advocate Medical Group
Locations (3):
- United States (3):
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Edward Hospital, Naperville, Illinois